CLINICAL TRIAL: NCT01697241
Title: The Effect of Education and Supervised Exercise vs. Education Alone on Time to Total Hip Replacement in Patients With Hip Osteoarthritis Considered Eligible for Surgery
Brief Title: Effect of Exercise as Non-surgical Treatments on Time to Total Hip Replacement Surgery
Acronym: HipSPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Institute for Clinical Research, Denmark (Industry); Vejle Hospital (Other); Region of Southern Denmark (Other); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Carsten Jensen, Assistant Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20120109
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis
Keywords: Exercise Therapy; Education; Osteoarthritis; Hip; Hip replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised exercise and patient education (Experimental): The entire duration of the intervention is 12 weeks, and consists of 24 sessions each lasting 60-70 minutes. Patients will receive two types of exercises, delivered on separate days. One type of exercise is individualized, goal-based neuromuscular training (NEMEX) in groups with progression guided by the patient's neuromuscular function (12 sessions). The other type of exercise is individualized, intensive resistance training (RT) in groups with each exercise progression guided by load (12 sessions).
  Interventions: Other: Supervised exercise; Other: Patient education
- Patient Education (Other): The patient education program is designed to educate the patients about hip OA during 3 sessions of 90 min. duration
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Supervised exercise — Patients in the exercise groups will receive two types of exercise, delivered on separate days. One type of exercise is individualized, goal-based neuromuscular training (NEMEX-TJR) in groups with progression guided by the patient's neuromuscular function. The other type of exercise is individualized, intensive resistance training (RT) in groups with each exercise progression guided by load. Each of the two types of exercise will be offered weekly during the 12 week intervention period in sessions lasting 60-70 minutes. Thus, the entire exercise intervention consists of 24 sessions
  Other Names: NEMEX-TJR and RT
  Arms: Supervised exercise and patient education
Other: Patient education — The patient education program is designed to educate the patients about hip osteoarthritis during 3 sessions of 90 min. duration
  Other Names: BOA

SUMMARY:
The aim of this trial is to test the hypothesis that patients with severe hip osteoarthritis postpone time to hip replacement surgery following participation in a patient education and supervised exercise program when compared to patients receiving patient education alone.

DETAILED DESCRIPTION:
Hip replacements are performed at an increasing rate, also in younger and less disabled patients. Recent studies indicate non-surgical interventions being effective in reducing pain and disability also at later stages of disease when hip replacement is considered. Possible, non-surgical treatments can be used to postpone hip replacement. The effect of education and supervised exercise on time to hip replacement is largely unknown

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older
* Indication for total hip arthroplasty
* Residency within local municipal or willing to commute

Exclusion Criteria:

* Inflammatory joint disease
* Earlier ipsilateral proximal femur fracture
* Hip pain < 3 months
* Neuropathy or neuromuscular disease
* Malignant disease
* Diseases where a moderate level of physical exercise is contraindicated
* Unable to speak or read Danish
* Unable to participate for other reasons
* Refuse to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cumulative Survival analysis (Kaplan-Maier survival curve) | one year
  Cumulative Survival analysis as time in days without surgery since inclusion

SECONDARY OUTCOMES:
The Hip disability and Osteoarthritis Outcome Score (HOOS 2.0) | Baseline, 3 and 12 months
  HOOS is patient-reported outcome measure with 5 subscales for pain, other symptoms, function in daily living, function in sport and recreation and hip related Quality of Life. A 5-point Likert-scale is used and converted into a 100-point scale with zero indicating the worst possible health (http://www.koos.nu).
University of California Los Angeles activity score (UCLA) | Baseline, 3 and 12 months
  Physical activity levels in populations. UCLA is a 10-point likert scale recommended and used extensively in similar populations
Global perceived effect (GPE) score | 3 and 12 months
  Patients will be asked to rate possible change in their pain, symptoms, ADL, sports and recreation, quality of life, level of physical activity since the initial administration (baseline) on a 7-point Likert-scale.

OTHER OUTCOMES:
Self-reported exercise pain (VAS-scale) | 3 months
  Pain intensity using the VAS-scale. Participants will be followed for the duration of the exercise intervention (3 months) and be asked to rate pain intensity before and after each exercise session (total 24 sessions)
Exercise adherence | 3 months
  'The extent to which a person's behavior corresponds with agreed recommendations from a health care provider' using no. of weeks, and no. of completed sessions
Cost-effectiveness analysis | 12 months
  Cost-effectiveness analysis will be estimated as the ratio between cost of the intervention and the effect it produces. The total cost will be estimated from register-based costing of primary care, secondary care and patient's out-of-pocket costs (transportation expenses and time spent on transportation and receiving health care). Patient-reported values are weighted using Danish tariffs
General health status EuroQol (EQ-5D-5L) | Baseline, 3 and 12 months
  The EQ-5D is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression (http://www.euroqol.org)
Mechanical Muscle Function | Baseline, 3 and 12 months
  Isometric muscle strength (iMVC) will be collected for knee extensors, hip extensors, -flexors and hip abductors.
Physical performance battery | Baseline, 3 and 12 months
  Physical performance-based measures will include; 30 s chair stand (number completed), 20 meter fast-paced walk (time in (s)), 30 s single-leg knee bending (number completed), and timed up and go (time in sec.)
Poor compliance | 3 months
  Reasons for poor compliance will be recorded.
Joint specific adverse events | 3 months
  Joint specific adverse events will be determined as: 1) not attending a training session and/or ceasing training because of increased pain/problems in the index joint related to the training; and 2) self-reported exercise pain > 5 on the VAS-scale after training. The reasons for not attending a session due to pain/problems related to training or to other reasons will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Jensen, PhD, Principal Investigator — Orthopedic Research Unit, Dept. of Orthopedic Surgery and Traumatology, Odense University Hospital, Denmark. Institute of Clinical Research, University of Southern Denmark, Denmark
Locations (2):
- Denmark (2):
  - Dept. of Orthopedic Surgery and Traumatology, Odense University Hospital, Denmark, Odense
  - Sector for Hip and Knee Replacement, Dept. of Orthopaedics, Vejle Hospital, Denmark, Vejle

REFERENCES:
- [Derived] Jensen C, Roos EM, Kjaersgaard-Andersen P, Overgaard S. The effect of education and supervised exercise vs. education alone on the time to total hip replacement in patients with severe hip osteoarthritis. A randomized clinical trial protocol. BMC Musculoskelet Disord. 2013 Jan 14;14:21. doi: 10.1186/1471-2474-14-21. PMID 23311889